CLINICAL TRIAL: NCT00592371
Title: Head and Neck Cancer Screening and Serum Repository
Status: Completed | Type: Observational
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: 59102
Record Dates: First submitted 2007-12-27; First posted 2008-01-14 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-09

CONDITIONS: Head and Neck Squamous Cell Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

SUMMARY:
Head and Neck Squaumous Cell Cancer(HNSCC) is the 6th most common cancer in the United States and the 3rd most common worldwide. Risk factors include abuse to tobacco and alcohol. Survival is related to stage of HNSCC when treatment is sought. Most HNSCC patients present with advanced staged disease. This screening activity will educate patients with HNSCC rick factors and screen for pre malignant and/or early staged lesions.

DETAILED DESCRIPTION:
Otolaryngology staff memebers and residents will perform head and neck examinations upon participants after the participant has completed their questionnaire and had the opportunity to partcipate in the research portion by having blood drawn. A suspicious head and neck examination will be considered abnormal, and further recommendations for follow-up will be made. Participants will be provided with a list of practicing head and neck surgeons within the state of Arkansas.

ELIGIBILITY:
Inclusion Criteria:

Exclusion Criteria:

* Under the age of 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2006-03; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brendan Stack, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States